CLINICAL TRIAL: NCT04585828
Title: Comparison of Double Pad Fiber Optic Device Versus Conventional Phototherapy for Treatment of Neonatal Hyperbilirubinemia
Brief Title: Comparison of Double Pad Fiber Optic Device Versus Conventional Phototherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71051
Record Dates: First submitted 2020-09-21; First posted 2020-10-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bili Cocoon (Experimental): The infants will be treated with phototherapy using a double sided fiber optic pad called Bili Cocoon with an irradiance of 30 uW/cm2/nm from both sides.
  Interventions: Device: Phototherapy with double sided fiber optic pads with blue light at irradiance 30 uW/cm2/nm using Bili Cocoon
- Conventional blue light (Active Comparator): The infants will be treated with blue light from above at 30 Uw/cm2/nm which is the standard treatment.
  Interventions: Device: Phototherapy from above using NeoBlue at irradiance of 30 uW/cm2/nm

INTERVENTIONS:
Device: Phototherapy with double sided fiber optic pads with blue light at irradiance 30 uW/cm2/nm using Bili Cocoon — The baby will be treated with Bilicocoon for 24 hours. Decrease of total serum biliurubin will be evalueated hereafter.
  Arms: Bili Cocoon
Device: Phototherapy from above using NeoBlue at irradiance of 30 uW/cm2/nm — The baby will be treated with phototherapy from above for 24 hours. Decrease of total serum bilirubin will be evaluated hereafter.
  Arms: Conventional blue light

SUMMARY:
A randomized study of phototherapy for neonatal hyperbilirubinemia. The intervention group is treated with a double pad fiber optic device and the control group with conventional blue ligt phototherapy from above. Both treatments are well known and used. The primary outcome is to explore the parents experience with the two different treatment modalities by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal icterus and total serum bilirubin above threshold for phototherapy.
* Gestational age ≥ 33 weeks
* Birth weight ≥ 1800 gr
* Postnatal age > 24 hours and < 2 weeks

Exclusion Criteria:

* Hemolysis due to isoimmunization
* Very high or rapidly rising total serum bilirubin

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Questionnaire on the parents experience with the phototherapy treatment | Day 1 of phototherapy
  Parents experience of phototherapy.
  Questions at time of beginning phototherapy (1):
  "What did you feel at the time your baby started treatment with phototherapy?"
  Questions after phototherapy (2):
  "What did you experience with your baby during the time of phototherapy?"
  The parents answer on a scale from "I agree, I partly agree, N/A, I partly disagreee, I disagree"
  Examples of questions:
  "I felt well informed about the indication and use of phototherapy" (Answer: I agree, partly agree, disagreee etc,)
  "I was difficult to breastfeed while my baby was on phototherapy" (Answer as above described)

SECONDARY OUTCOMES:
Effect of phototherapy | Measurement of bilirubin before phototherapy and after 24 hours
  Change in total serum bilirubin